CLINICAL TRIAL: NCT05750836
Title: Assessment and Prevention of Caregiver Burden in Oncology
Acronym: PREPAC-01
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ICO-2022-03
Record Dates: First submitted 2023-02-20; First posted 2023-03-02 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-02

CONDITIONS: Oncology; Caregiver Burden
Keywords: Nurse; Supportive Care; Zarit scale; Caregiver Burden
MeSH Terms: conditions — Neoplasms; Caregiver Burden

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Specific nursing support (Experimental): The caregivers benefit from specific nursing support.
  Interventions: Other: Specific nursing support
- No specific nursing support (Active Comparator): Caregivers do not receive any specific support from the nurses.
  Interventions: Other: Non-specific nursing support

INTERVENTIONS:
Other: Specific nursing support — * 3 mandatory on-site nursing consultations with the patient's caregiver at inclusion, 6 months and 12 months post-randomisation.The caregivers will complete the questionnaires (Zarit scale, Hospital Anxiety and Depression scale, Medical Outcome Study Short Form - 36, Caregiver's satisfaction).
  * interviews once a month with a nurse either by phone, on-site consultation or teleconsultation.
  Nurses assess the general health of the caregiver and Identify the socio-professional situation of the caregiver
  Arms: Specific nursing support
Other: Non-specific nursing support — Caregivers will only have to complete on site Health indicators, Zarit scale, Hospital Anxiety and Depression scale, Medical Outcome Study Short Form - 36 at inclusion, 6 months and 12 months post-randomisation.
  Arms: No specific nursing support

SUMMARY:
The goal of this randomized, open and controlled supportive care study is to see if we can reduce the burden on the caregiver by offering the caregiver systematic and regular support from the nurse (APN, nurse coordinator in French health care organisations) compared to a support focused on the patient. At the same time, we will also evaluate the impact of this personalised support for the caregiver on their anxiety and quality of life.

Participants will caregivers of a patient who started a line (any line) of systemic treatment for a solid tumour since less than 3 months or in an active palliative situation since less than 1 month.

Researchers will compare 2 groups : a group where caregivers benefit from specific nursing support and a group of caregivers with no specific nursing support.

The specific support includes 3 mandatory on-site nursing consultations with the patient's caregiver and interviews once a month with a nurse either by phone, on-site consultation or teleconsultation.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver designated by the patient;
* Caregiver of a patient who started a line (any line) of systemic treatment for a solid tumour since less than 3 months or in an active palliative situation since less than 1 month;
* Caregiver of patient already cared for by a nurse before inclusion or going to start a nursing follow-up;
* Caregiver of a patient with a score ≥2 of social fragility and/or psychological fragility and/or nutritional fragility and/or complexity;

Exclusion Criteria:

* Patient whose life expectancy is assumed to be < 6 months;
* Patient living in an institution (EHPAD, MAS, SSR, MCO, USLD) at inclusion;
* Caregiver declared as having a pathology that could alter his/her capacity to support (psychiatric history, dementia…) or under guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Caregiver burden | at 6 months post-randomisation
  Comparison in the 2 groups. Burden score is assessed using the ZARIT SCALE. The test consists of 22 questions that the caregiver has to score from 0 to 4, the whole giving a score from 0 to 88. 0 means no burden, 88 means that the burden is severe

SECONDARY OUTCOMES:
The level of anxiety/depression of the caregiver | at month 6 (M6) and month 12 (M12) post-randomisation.
  Comparaison in the 2 groups.
  Hospital Anxiety and Depression scale consists of 14 items to which participants respond on a 4-point Likert scale. Seven items assess anxiety and seven items assess depression. Anxiety and depression scores can range from 0 (no symptoms) to 21 (significant presence of symptoms). Threshold scores were determined as follows:
  * between 0 and 7 : no symptoms of anxiety or depression;
  * between 8 and 10 : some moderate symptoms (mild anxiety or depression);
  * score of 11 or more : significant number of symptoms (severe anxiety or depression).
Caregiver's quality of life | at month 6 (M6) and month 12 (M12) post-randomisation.
  Comparison in the 2 groups. The generic self-questionnaire SF36 consists of 36 items concerning the last four weeks before the test and divided into 8 dimensions (Physical activity ; Life and relationships with others ; Physical pain; Perceived health ; Vitality; Limitations due to the psychological state; Limitations due to the physical state; Psychological health).
  These eight dimensions are used to measure two summary scores of the quality of life of individuals: the physical composite score (PCS) and the mental composite score (MCS). (score from 0 to 100).
  A low score reflects a perception of poor health, loss of function, presence of pain. A high score reflects a perception of good health, absence of functional deficit and pain.
Caregiver's satisfaction | at month 6 (M6) and month 12 (M12) post-randomisation.
  Only arm B. P-GIC questionnaire consists of a single question asking the caregiver about their overall impression of change in specific support care. The caregiver is given the following 8 options and asked to indicate which of these best describes the perceived change: I don't know, Very strongly positive, Strongly positive, Slightly positive, No change, Slightly negative, Strongly negative, Very strongly negative.

CONTACTS AND LOCATIONS:
Overall Officials: Céline THOMAS, Nurse, Principal Investigator — Institut de Cancérologie de l'Ouest
Locations (5):
- France (5):
  - CH Cholet, Cholet
  - Centre Antoine Lacassagne, Nice
  - Centre Henri Bequerel, Rouen
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - CH Mémorial de Saint Lo, Saint-Lô